CLINICAL TRIAL: NCT03800056
Title: Characterization of the Fungal Origins in the Autoimmune Polyendocrinopathy of Type 1 Compared With the Autoimmune Polyendocrinopathies of Type 2
Acronym: APECED2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_36; 2017-A03135-48 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Polyendocrinopathies, Autoimmune
Keywords: APECED syndrome; autoimmune polyendocrinopathy; chronic mucocutaneous candidiasis
MeSH Terms: conditions — Polyendocrinopathies, Autoimmune; Candidiasis, Chronic Mucocutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 2x7mL EDTA tubes and 1x7 mL dry tube for the collection of DNA, plasma ans serum.
  * a urine sample and an oral collection for the characterization of fungal flora
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 APS 1: Patients with a APS type 1 whose molecular diagnosis (mutation of the AIRE gene) has been established in the diagnosis of the disease, regardless of their mycological status (history of mycosis) or the presence of antifungal treatment.
- Group 2 APS2: Patients with APS type 2: - with adrenal insufficiency for 50% of them. - a delay of two weeks after stopping antifungal or antibiotic treatment in patients is to be respected.

SUMMARY:
Autoimmune polyendocrinopathy candidiasis ectodermal dystrophy (APECED) is an autosomal recessive disease caused by mutations in the autoimmune regulator (AIRE) gene, characterized by the clinical triad of chronic mucocutaneous candidiasis (CMC), hypoparathyroidism, and adrenal insufficiency. CMC can be complicated by systemic candidiasis or oral squamous cell carcinomas (SCCs) and may lead to death. The role of chronic Candida infection in the etiopathogenesis of oral SCC is unclear. Long term use of fluconazole lead to emergence of C. albicans strains with azoles decreased susceptibility. CMC is associated with an impaired Th17 cell response, however, it remains unclear whether decreased serum IL-17 and IL-22 levels are related to a defect in cytokine production or to neutralizing autoantibodies resulting from mutations in the AIRE gene

ELIGIBILITY:
Inclusion Criteria:

1. For both of groups, inclusion criteria are :

   * children aged 0 to 17 years old with the consent of both parents, and men and women between the ages of 18 and 85.
   * a reasonable delay of 2 weeks after the resolution of an intercurrent infectious episode is to be observed.
   * assent of the patient after information adapted to his age and his degree of understanding.
   * informed, express and written consent of the patient or of each of the holders of parental authority.
2. Inclusion criteria specific to group 1: Patients with a APS type 1 whose molecular diagnosis (mutation of the AIRE gene) has been established in the diagnosis of the disease, regardless of their mycological status (history of mycosis) or the presence of antifungal treatment.
3. Inclusion criteria specific to group 2 : Patients with APS type 2: - with adrenal insufficiency for 50% of them. - a delay of two weeks after stopping antifungal or antibiotic treatment in patients is to be respected.

Exclusion Criteria:

* impossibility to receive informed information for adults, or impossibility to receive enlightened information for the holders of parental authority if minor subject
* inability to participate in the entire study, refusal to sign the consent.
* people in an emergency situation.
* persons deprived of their liberty.
* pregnant or lactating woman (pregnant women will be offered to participate in the study after delivery).

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be included during their routine follow-up for adrenal insufficiency or hypoparathyroidism in the endocrinology department of the University Hospital of Lille, in adult or pediatric endocrinology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
the frequency of appearance of Candida yeast strains | Baseline: one session
  the frequency of appearance of Candida yeast strains found in mycological samples from both urinary and oral patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine VANTYGHEM, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France